CLINICAL TRIAL: NCT06378983
Title: A Single Center, Prospective Randomized Controlled Clinical Trial on the Efficacy and Safety of Microneedle Radiofrequency Combined With Oral Isotretinoin in Moderate to Severe Acne Vulgaris
Brief Title: Clinical Trial of Microneedle Radiofrequency Combined With Oral Isotretinoin in Moderate to Severe Acne
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SYSKY-2023-1149-02
Record Dates: First submitted 2024-02-20; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Moderate to Severe Acne Vulgaris
Keywords: microneedle radiofrequency; isotretinoin; acne vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Isotretinoin; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- oral isotretinoin combined with microneedle radiofrequency therapy group (Experimental): Oral isotretinoin was administered using the same method as the isotretinoin group, while microneedle radiofrequency therapy was also administered.Using the Peninsula radiofrequency therapy device (Peninsula Company, China). A total of 3 treatments were conducted, with a treatment interval of 1 month, and the total course of treatment was 8 weeks.
  Interventions: Other: Oral isotretinoin combined with microneedle radiofrequency therapy
- oral isotretinoin alone group (Other): Oral isotretinoin capsules at a dose of 10mg/time, once per day, orally, for a total course of 8 weeks.
  Interventions: Drug: Oral isotretinoin

INTERVENTIONS:
Drug: Oral isotretinoin — Oral isotretinoin
  Other Names: Control group
  Arms: oral isotretinoin alone group
Other: Oral isotretinoin combined with microneedle radiofrequency therapy — Oral isotretinoin combined with microneedle radiofrequency therapy
  Other Names: Experimental group
  Arms: oral isotretinoin combined with microneedle radiofrequency therapy group

SUMMARY:
This study plans to select 100 AV patients and randomly divide them into two groups in a 1:1 ratio: the experimental group will be treated with MRF combined with oral isotretinoic acid for 8 consecutive weeks, with a total of 3 MRF treatments at weeks 1, 4, and 8. The control group received oral administration of isotretinoic acid alone for 8 weeks. The main observation indicators are the percentage of effective skin injury clearance achieved by subjects at week 20, as well as the change in ECCA acne scar score compared to baseline at week 20. I hope this study can clarify that the combination therapy of the two can achieve the effects of improving efficacy, shortening treatment course, reducing recurrence, not increasing adverse reactions, and reducing the risk of scar formation.

DETAILED DESCRIPTION:
Acne vulgaris (AV) is a chronic inflammatory skin disease that is prone to damage during adolescence. Based on the damage to appearance, it has a negative impact on the psychological and daily life of AV patients, increasing their economic burden. Isoretinoic acid is currently an oral medication targeting the four key pathological and physiological stages of AV, but adverse reactions are common, safe and effective, and the treatment or drug letter that can prevent scar formation remains unclear. Our preliminary research has confirmed that microneedle radiofrequency therapy (MRF) can effectively treat AV and improve post AV pigmentation and scar formation. To further confirm the efficacy and safety of MRF combined with oral isotretinoic acid in the treatment of moderate to severe AV, we plan to conduct a randomized, oral controlled prospective clinical study. This study plans to select 100 AV patients and randomly assign them to two groups in a 1:1 ratio: the experimental group was treated with MRF combined with oral isotretinoin for 8 weeks of continuous oral medication, and a total of 3 MRF sessions were conducted at weeks 1, 4, and 8. The control group was treated with oral isotretinoin alone for 8 weeks. The main observation indicators are the percentage of effective skin lesion clearance rate achieved by subjects at week 20, as well as the change in ECCA acne scar score from baseline at week 20. It is hoped that this study can clarify that the combination therapy of the two can achieve the effects of improving efficacy, shortening treatment course, reducing recurrence, not increasing adverse reactions, and reducing the risk of scar formation.

ELIGIBILITY:
Inclusion Criteria:

1. Provide a signed and dated informed consent form before conducting any research related processes
2. Male and female aged 14-65
3. Patients clinically diagnosed with moderate to severe acne vulgaris (according to the Chinese Acne Treatment Guidelines, revised in 2019) must meet the Pillsbury International Modified Classification (see Appendix 5), which belongs to level II-III, and the IGA (Investigator Global Assessment) assessed by the study physician as moderate (3) or severe (4)
4. Type III-IV skin according to Fitzpatrick scale
5. Adhere to all lifestyle precautions throughout the entire study period and refrain from using other acne treatment drugs, etc.

Exclusion Criteria:

1. Pregnant women or women planning to conceive during the study period, pregnant or lactating women, and fertile female subjects who are unable to use or do not plan to use medically acceptable contraceptive measures. Male subjects who do not plan to use medically acceptable contraceptive measures.
2. For women with fertility: did not use medically approved contraceptive measures for at least one month prior to screening, and did not agree to use medically approved contraceptive measures during the study period or within 30 days after the end of study drug use.
3. Individuals who currently meet any of the following conditions in clinical practice: aggregate acne, fulminant acne, secondary acne (drug-induced acne), or any facial skin condition or facial hair that may interfere with clinical evaluation (such as sideburns, sideburns, beard). The following types of skin diseases that can interfere with the evaluation of acne vulgaris include folliculitis, rosacea, demodex, pustular vasculitis, mechanical acne, occupational acne including oily or tar acne, as well as chloroacne, facial disseminated lupus lesions, etc.
4. Facial sunburn
5. Researchers believe that laboratory values or electrocardiogram examinations with clinically significant abnormalities should be screened, including but not limited to the following situations (if the screening period test results are difficult to explain, according to the researcher's judgment, a repeated measurement is allowed): 1) Fasting blood glucose is greater than the upper limit of normal values; 2) Creatine kinase is greater than or equal to twice the upper limit of normal value; 3) Liver function (AST or ALT) greater than 1.5 times the upper limit of normal value; 4) Creatinine is higher than the upper limit of normal value; 5) Female pregnancy test positive; 6) Abnormal ECG examination has clinical significance.
6. Participated in clinical studies of other drugs and devices within the first three months of screening;
7. Select subjects who have undergone major surgery (i.e. require general anesthesia) within the first 12 weeks, have not fully recovered from surgery, or are expected to undergo surgery during the study period.
8. Subjects with any of the following medical histories should be excluded: 1) those who are allergic to isotretinoids or any component of the investigational drug, or have a history of multiple drug allergies; 2) known or suspected precancerous lesions or malignant diseases, including a history of malignant tumors within the previous 5 years of screening (such as evidence of any tumor activity within the past 5 years, or diagnosed with malignant tumors within that period, excludingSkin cancer treated with Gong therapy.
9. Subjects who have used any of the following drugs before enrollment in the study, or who are currently using these drugs and have not completed the washout period as required below: Note: The washout period should be calculated from the expected randomization date (day 0). The random allocation date can be adjusted to ensure that the subjects complete the washout period.1) Within one week before randomization: all medical skincare products with acne relieving effects; 2) Within 2 weeks before randomization: topical acne treatment drugs, including but not limited to: topical corticosteroids; External use of retinoic acid drugs; Topical application of benzoyl peroxide; Topical antibiotics (clindamycin; erythromycin; lincomycin, etc.); External use of azelaic acid drugs; 3) Within the first 4 weeks of randomization: laser and photodynamic therapy; Antibiotics used throughout the body (tetracyclines, macrolides, etc.); Finasteride; Systemic use of sex hormones (estrogen, progesterone, and progesterone); Chinese medicine or traditional Chinese patent medicines and simple preparations for acne treatment; Immunosuppressants (cyclosporine/Tripterygium wilfordii/Methotrexate, etc.); Immunomodulators (glycyrrhizic acid glycoside/tanshinone/berberine, etc.) 4) Within the first 12 weeks of randomization: systemic administration of isotretinoids; Use corticosteroids throughout the body; Biological agents with immunomodulatory effects, such as omalizumab.
10. Subjects with severe liver, kidney, cardiovascular, respiratory, endocrine, hematological, urinary, metabolic, central nervous system, or autoimmune diseases.
11. Screening shows a history of drug abuse and alcohol abuse within the first 2 years.
12. The research center personnel and/or their immediate family members who directly participated in this study. Immediate relatives refer to spouses, parents, children or siblings (who are related by blood or legally adopted).
13. Other situations that the researcher deems unsuitable for participation in the study.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in ECCA acne scar score from baseline at week 20 | week 20
  Two experienced dermatologists who are in a blind state will evaluate the patient's ECCA score. If the results are inconsistent, the third evaluator will evaluate and serve as the final result.
The percentage of effective skin lesion clearance rate in the 20th week | week 20
  Two experienced dermatologists who are in a blind state will perform facial skin lesion counting on the patient. If the results are inconsistent, the third evaluator will evaluate and serve as the final result.

CONTACTS AND LOCATIONS:
Overall Officials: Sha Lu, Study Director — Department of Dermatology, Sun Yat-sen Memorial Hospital, Sun Yat-Sen University
Locations (1):
- Department of Dermatology and Venereology, Sun Yat-sen Memorial Hospital, Sun Yat-sen University., Guangzhou, China